CLINICAL TRIAL: NCT04196608
Title: In Vitro Activity of Ceftolozane/Tazobactam and Imipenem/Relebactam in Clinical Isolates of Pseudomonas Aeruginosa and Enterobacterales Collected From Hematology and Oncology Patients
Acronym: ACTHEON
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emilio Bouza (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Emilio Bouza, Phd, MD Senior Assesor, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: MICRO.HGUGM.2019-008
Record Dates: First submitted 2019-12-03; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Ceftolozane/Tazobactam; Imipenem/Relebactam; Hematology and Oncology
MeSH Terms: conditions — Neoplasms | interventions — ceftolozane, tazobactam drug combination; imipenem, cilastatin and relebactam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- P. aeruginosa isolates: All isolates will be sent to the Central Laboratory, where identification will be confirmed by MALDI-TOF and susceptibility testing against ceftolozane/tazobactam, imipenem- relebactam and comparative agents will be performed
  Interventions: Drug: Ceftolozane/tazobactam; Drug: imipenem- relebactam
- Enterobacterales isolates: All isolates will be sent to the Central Laboratory, where identification will be confirmed by MALDI-TOF and susceptibility testing against ceftolozane/tazobactam, imipenem- relebactam and comparative agents will be performed
  Interventions: Drug: Ceftolozane/tazobactam; Drug: imipenem- relebactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — Minimum inhibitory concentrations (MICs) will be determined by the standard broth microdilution method (standard ISO method 20776-1:2006) using dry-form Sensititre panels (Thermo Fisher Scientific, Denmark) and will be interpreted according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) and the Clinical and Laboratory Standards Institute (CLSI) criteria
Drug: imipenem- relebactam — Minimum inhibitory concentrations (MICs) will be determined by the standard broth microdilution method (standard ISO method 20776-1:2006) using dry-form Sensititre panels (Thermo Fisher Scientific, Denmark) and will be interpreted according to the European Committee on Antimicrobial Susceptibility Testing (EUCAST) and the Clinical and Laboratory Standards Institute (CLSI) criteria

SUMMARY:
The purpose of the ACTHEON Study is to evaluate the in vitro activity of ceftolozane-tazobactam, imipenem-relebactam and comparator agents (amoxicillin- clavulanate, piperacillin-tazobactam, ceftazidime, cefotaxime, cefepime, imipenem, meropenem, levofloxacin and amikacin; see list more details on page 7) against clinical isolates of P. aeruginosa and Enterobacterales prospectively collected from hematology and oncology patients with complicated intra-abdominal infections (cIAIs), complicated urinary infections (cUTIs), lower respiratory tract infections (LRTIs), and blood stream infections (BSIs) from 15 participating centers in Spain

ELIGIBILITY:
Inclusion Criteria:

* P. aeruginosa isolates
* Enterobacterales isolates

Exclusion Criteria:

* Non P. aeruginosa isolates
* Non Enterobacterales isolates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating laboratories will prospectively collect the first 1,005 clinical isolates (510 P. aeruginosa isolates and 495 Enterobacterales isolates) starting in a preestablished date from patients with cIAIs, cUTIs, LRTIs, or BSIs
Sampling Method: Non-Probability Sample
Enrollment: 1005 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Summary MIC and its distributions as susceptible, intermediate and resistant | 31 october 2020
  Summary of MIC data, distribution presented as the cumulative MIC frequency, MIC50, MIC90, and MIC range for each antimicrobial and species.
Summary of percentages of isolates | 31 october 2020
  Summary of percentages of isolates interpreted as susceptible, intermediate and resistant isolates according to CLSI and EUCAST guidelines, when available, for each species and for the total study isolates.

CONTACTS AND LOCATIONS:
Locations (1):
- HG Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Fiveteen laboratories (Participating laboratories) will participate under the direction of Dr. E. Cercenado, Department of Microbiology and Infectious Diseases, Gregorio Marañón University Hospital, Madrid, Spain (Central laboratory), on behalf of the GEIRAS-SEIMC (Group for the Study of Healthcare-Related Infections of the Spanish Society for Infectious Diseases and Clinical Microbiology).